CLINICAL TRIAL: NCT01782586
Title: Multicenter Validation of Gene Expression Markers of Renal Allograft Functional Decline (GEN-04)
Brief Title: Validation of Gene Expression Markers of Renal Allograft Functional Decline
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genomics of Transplantation Cooperative Research Program (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAIT GEN-04
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Kidney Transplant Recipients
Keywords: kidney transplant; gene expression markers; renal allograft function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1-year surveillance biopsy and blood on 494 conventional kidney transplant participants from the 4 participating sites.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if certain genes found in a kidney biopsy performed at one-year post transplant can predict which transplanted kidneys will have decreased kidney function within five years post-transplant.

DETAILED DESCRIPTION:
Gene expression profiling is used to study the activity of genes. Each gene has an "on/off" switch that controls how they are expressed in a cell, as well as a "volume control" that increases or decreases the level of expression of a particular gene as necessary. Researchers want to see if the presence and abundance of certain transcripts in a kidney biopsy at one year after transplant can predict which kidneys will have reduced function over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) conventional renal transplant recipient.
* Patients who have given informed consent and are willing to comply with the protocol.

Exclusion Criteria:

* ABO incompatible kidney transplants.
* Positive crossmatch kidney transplants (T cell crossmatch >100, B flow cytometric crossmatch >150).
* Simultaneous kidney and extra-renal organ transplants including pancreas, liver, heart, lung, etc. Subjects who had previous extra renal transplants may be included in the study.
* Patients taking chronic anticoagulation, which includes Coumadin, Plavix and any type of heparin. Aspirin is acceptable but must be stopped 5 days prior to the renal biopsy.
* An inability to have the 1-year renal biopsy performed within the acceptable protocol window (Months 11-14 [Days 301-420] post-transplant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Renal Function Decline | Baseline to 1 year
  The primary endpoint for this study is defined as a progressive decline in renal function in participants with good function at 1 year. These "Progressors" are defined by all of the following criteria:
  1. 1 year estimated GFR (eGFR) by MDRD equation of >40 ml/min.
  2. Decline in eGFR beyond 1 year during the time frame of this study (minimum 2.6 years after transplant and up to 5 years after transplant) with a slope of <-6.1% (i.e. slope of decline of renal function is >6.1%).
  3. >20% decline in eGFR from 1 year post-transplant to latest follow-up point.
  4. At least one eGFR (MDRD) interval < 60 ml/min.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Stegall, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (4):
- United States (4):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait